CLINICAL TRIAL: NCT03055065
Title: Epidemiological, Prospective, Multicentric, Open Study To Assess The Characteristics And Frequency Of Adenoviral Conjunctivitis As Diagnosed With The Point Of Care AdenoPlus® Test In Patients Suffering From Acute Conjunctivitis
Brief Title: ADenoVirus Initiative Study in Epidemiology in Italy
Status: Completed | Type: Observational
Sponsor: NicOx (Industry)
Responsible Party: Sponsor
Other Study IDs: ADVISE Italy
Record Dates: First submitted 2014-09-29; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Viral Conjunctivitis
Keywords: Adenoviral conjunctivitis diagnosed with AdenoPlus™ Test
MeSH Terms: conditions — Conjunctivitis, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study is to assess the characteristics and frequency of adenovirus conjunctivitis in a population of male and female patients from one year of age who present signs and symptoms of acute conjunctivitis.

DETAILED DESCRIPTION:
Epidemiological, prospective, open, multicentric trial in patients suffering from acute conjunctivitis who will undergo a rapid diagnostic test for adenoviral conjunctivitis at the time of their visit to the ophthalmologist office, at the emergency room or during hospitalization. This epidemiological study will include approximately 500 patients in Italy. The planned duration of the study is one year from the first patient visit to the last patient visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients of at least one year of age presenting acute (for less than 7 days) conjunctivitis signs and symptoms.
* Patient or / and legal representative (if patient below 18 years of age) must be able to provide oral consent for the collection and treatment of the questionnaire data.
* No history of hypersensitivity to corn starch, talcum powder or Dacron (sampling fleece components).

Exclusion Criteria:

* Current use or having received (within the last 7 days) local antiviral therapies such as povidone iodine or ganciclovir, or topical steroids or immunomodulators such as cyclosporine which may interfere with the test result.
* Previous enrolment in the present study.
* Any direct involvement with the study conduct at site or any family link with study site staff.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any female and male patients from one year of age with signs and symptoms of acute conjunctivitis either seen during ophthalmology consultations or who are in the emergency room or hospitalized, can be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with adenovirus conjunctivitis | During the visit to the ophthalmologist (one visit)
  The percentage of patients with adenovirus conjunctivitis documented by a positive AdenoPlus® test over the tested population of male and female patients who present signs and symptoms of acute conjunctivitis.

OTHER OUTCOMES:
data collection: Seasonality and geographic repartition observed. | One day during the visit to the ophthalmologist before and just after the AdenoPlus® test done on the same day (one visit)
  The number of patients with adenovirus conjunctivitis who visited the ophthalmologist in spring, summer, autumn and winter and their geographic area (e.g. by hospital, by area).
Percentage of each eye signs and symptoms measured by questionnaire | One day during the visit to the ophthalmologist before and just after the AdenoPlus® test done on the same day (one visit)
  The percentage of each eye signs and symptoms for both the patients with positive and negative AdenoPlus® tests
Duration of the disease measured by questionnaire | One day during the visit to the ophthalmologist before and just after the AdenoPlus® test done on the same day (one visit)
  the mean duration of the disease for both the patients with positive and negative AdenoPlus® tests
Number of follow-up visits done measured by questionnaire | One day during the visit to the ophthalmologist before and just after the AdenoPlus® test done on the same day (one visit)
  The number or follow-up visit done
Diagnosis measured by questionnaire | One day during the visit to the ophthalmologist before and just after the AdenoPlus® test done on the same day (one visit)
  The correlation between the initial diagnosis (before AdenoPlus® test results) and the final diagnosis (post AdenoPlus® test results).
Resource utilization during the treatment | On day 1: at least once during the single visit to the ophthalmologist and if any also during the follow-up visit(s) at latest one year following visit 1
  Estimation of resource utilized during course of treatment (use of drugs, number of visits done by the patient…), .
Evaluation of the costs of resource utilization during the treatment | On day 1: at least once during the single visit to the ophthalmologist and if any also during the follow-up visit(s) at latest one year following visit 1
  associated costs of resources used during the treatment (use of drugs, number of visits done by the patient…), (which would be calculated by applying unit costs to resource use).
Patient/parent absenteeism linked to this disease measured by questionnaire | On day 1: at least once during the single visit to the ophthalmologist and if any also during the follow-up visit(s) at latest one year following visit 1
  Number of days out of work and/or out of school linked to this disease.
Safety assessment measured by data collection | On day 1: at least once during the single visit to the ophthalmologist and if any also during the follow-up visit(s) at latest one year following visit 1
  Number of adverse incidents (AIs) and events that are of significant (SEs) reported to Nicox

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fogagnolo, MD, Principal Investigator — Ospedale san Paolo Blocco
Locations (1):
- Clinica oculistica / Ospedale san Paolo, Milan, Italy